CLINICAL TRIAL: NCT04836143
Title: Eyes That Do Not Meet the Eligibility Criteria of Clinical Trials on Age-Related Macular Degeneration: Proportion of the Real-World Patient Population and Reasons for Exclusion
Status: Completed | Type: Observational
Sponsor: Kim's Eye Hospital (Other)
Responsible Party: Principal Investigator, Jae Hui Kim, Consultant, Kim's Eye Hospital
Other Study IDs: 2019-07-015
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Age-related Macular Degeneration
Keywords: Age-related Macular Degeneration; Polypoidal Choroidal Vasculopathy
MeSH Terms: conditions — Macular Degeneration; Polypoidal Choroidal Vasculopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Intravitreal anti-vascular endothelial growth factor injection — Intravitreal injection of either ranibizumab or aflibercept

SUMMARY:
The purpose of the present study was to evaluate the proportion of eyes that do not meet the eligibility criteria of clinical trials on neovascular AMD among the entire sample of eyes diagnosed with treatment-naïve neovascular AMD. The eligibility criteria of the VEGF Trap-Eye: Investigation of Efficacy and Safety in Wet AMD (VIEW) studies, were used for this investigation.

DETAILED DESCRIPTION:
Neovascular AMD is one of the primary causes of severe visual impairment in developed countries. Previously, laser photocoagulation or photodynamic therapy was used as its mainstay treatment. However, the efficacy of these treatment modalities has obvious limitations. In 2006, the FDA-approved anti-VEGF agent, ranibizumab, was introduced, followed by aflibercept in 2012. In addition, the off-label use of bevacizumab has been widely adopted. The introduction of these anti-VEGF agents has markedly improved the treatment outcomes of neovascular AMD, resulting in a significant decrease in the rate of visual loss and blindness. Currently, clinical trials are actively being performed to develop better treatment methods for neovascular AMD.

In general, conducting clinical trials are expensive and require years to complete. Therefore, estimating the time required to complete the planned patient enrollment is essential for establishing an efficient clinical trial plan. Clinical trials are usually conducted in a controlled environment and have sophisticated eligibility criteria. Thus, all patients cannot be enrolled into a trial, and some of them, or sometimes the majority of them, are excluded on the basis of the eligibility criteria.

Estimation of the proportion of patients in the study population who do not meet the eligibility criteria is important for several reasons. First, it may help to identify whether the results of the clinical trial can be applied to the real-world patients. Secondly, it may also help to predict the time required to finish the planned patient enrollment. In addition, if a particular set of criteria results in the exclusion of a relatively large number of patients, patient enrollment in future clinical trials could be accelerated by modifying some of these criteria. Furthermore, since the characteristics of neovascular AMD differ between Asian and Caucasian populations, obtaining data on Asian populations would be of great value.

Therefore, the purpose of the present study was to evaluate the proportion of eyes that do not meet the eligibility criteria of clinical trials on neovascular AMD among the entire sample of eyes diagnosed with treatment-naïve neovascular AMD. The eligibility criteria of the VEGF Trap-Eye: Investigation of Efficacy and Safety in Wet AMD (VIEW) studies, were used for this investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with treatment-naïve, active neovascular AMD between January 2017 and December 2017.
* Patients aged ≥ 50 years old
* Patients who received intravitreal anti-VEGF injection after the diagnosis

Exclusion Criteria:

- None

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with treatment-naive active neovascular AMD and were treated with anti-VEGF
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-01-26 (Actual); Study Completion 2020-07-26 (Actual)

PRIMARY OUTCOMES:
The proportion of eyes that do not meet the eligibility criteria of clinical trials on neovascular AMD among the entire sample of eyes diagnosed with treatment-naïve neovascular AMD | Baseline
  The proportion of eyes that do not meet the eligibility criteria of clinical trials on neovascular AMD among the entire sample of eyes diagnosed with treatment-naïve neovascular AMD. The eligibility criteria of the VEGF Trap-Eye: Investigation of Efficacy and Safety in Wet AMD (VIEW) studies, were used for this investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hui Kim, M.D., Principal Investigator — Kim's Eye Hospital, South Korea
Locations (1):
- Jae Hui Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Heier JS, Brown DM, Chong V, Korobelnik JF, Kaiser PK, Nguyen QD, Kirchhof B, Ho A, Ogura Y, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Soo Y, Anderesi M, Groetzbach G, Sommerauer B, Sandbrink R, Simader C, Schmidt-Erfurth U; VIEW 1 and VIEW 2 Study Groups. Intravitreal aflibercept (VEGF trap-eye) in wet age-related macular degeneration. Ophthalmology. 2012 Dec;119(12):2537-48. doi: 10.1016/j.ophtha.2012.09.006. Epub 2012 Oct 17. PMID 23084240
- [Result] Moore TJ, Zhang H, Anderson G, Alexander GC. Estimated Costs of Pivotal Trials for Novel Therapeutic Agents Approved by the US Food and Drug Administration, 2015-2016. JAMA Intern Med. 2018 Nov 1;178(11):1451-1457. doi: 10.1001/jamainternmed.2018.3931. PMID 30264133
- [Result] Sertkaya A, Wong HH, Jessup A, Beleche T. Key cost drivers of pharmaceutical clinical trials in the United States. Clin Trials. 2016 Apr;13(2):117-26. doi: 10.1177/1740774515625964. Epub 2016 Feb 8. PMID 26908540
- [Result] Kim JH, Chang YS, Kim JW, Kim CG, Lee DW. Age-related differences in the prevalence of subtypes of Neovascular age-related macular degeneration in the first diagnosed eye. Graefes Arch Clin Exp Ophthalmol. 2019 May;257(5):891-898. doi: 10.1007/s00417-018-04228-4. Epub 2019 Jan 7. PMID 30617580